CLINICAL TRIAL: NCT02194751
Title: Oncoquest-L Vaccine in Patients With Previously Untreated Stage III or IV, Asymptomatic, Non-bulky Follicular Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: XEME Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X13-21008
Record Dates: First submitted 2014-07-14; First posted 2014-07-18 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2020-07

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oncoquest-L vaccine (Experimental): Patients will receive a total of 5 single injections of Oncoquest-L; the first 2 doses administered will be separated by a 2-week interval and the remaining 3 doses will be administered each at 1-month intervals. With each dose of Oncoquest-L vaccine, the vaccine will be administered subcutaneously at 2 different sites in the upper arms or upper legs, with alternation of the injection sites with each administration.
  Interventions: Biological: Oncoquest-L vaccine

INTERVENTIONS:
Biological: Oncoquest-L vaccine — Patients will receive a total of 5 single administrations of Oncoquest-L; the first 2 doses administered will be separated by a 2-week interval and the remaining 3 doses will be administered each at 1-month intervals. With each dose of Oncoquest-L vaccine, the vaccine will be administered subcutaneously at 2 different sites in the upper arms or upper legs, with alternation of the injection sites with each administration. For each vaccination, a total of 1.0 mL of vaccine will be administered, divided into 2 subcutaneous injections of 0.5 mL each at 2 different injection sites.

SUMMARY:
This Phase II trial studies the overall tumor response of vaccine therapy in patientswith previously untreated Stage III or IV, asymptomatic, non-bulky follicular lymphoma. The vaccine contains an extract of the patient's own cancer cells and the immunostimulant protein, interleukin-2 (IL-2). It is hoped that when injected under the skin, the vaccine will enable the patient's immune system to recognize and destroy the cancer cells. The trial will also assess the safety of the vaccine, the time from vaccine treatment until the patient requires another type of anti-lymphoma treatment, progression-free survival, and the anti-tumor immune response.

DETAILED DESCRIPTION:
This is a single-arm open-label pilot Phase II study. Following informed consent, eligible subjects will undergo excisional biopsy of a lymphoma-containing lymph node for diagnosis and for generation of the Oncoquest-L vaccine. Patients will receive subcutaneous injections consisting of their autologous tumor-derived Oncoquest-L vaccine starting at approximately 4 to 8 weeks after the biopsy. The first two doses will be given at a 2-week interval and the remaining 3 doses at monthly intervals. Patients will be monitored for response by performing imaging studies at baseline and 1 month after the fifth vaccination (Week 19). Additional imaging studies will be performed every 3 months for the first year and every 6 months during the second year until relapse or disease progression whichever occurs sooner.

ELIGIBILITY:
Inclusion Criteria:

1. Follicular lymphoma (FL) grade 1, 2, or 3a diagnosed within 12 months of study enrollment
2. Age ≥ 18 years
3. Previously untreated Stage III or IV FL
4. A single peripheral lymph node of at least 1 x 1 cm in size accessible for excisional biopsy
5. Measurable or evaluable disease after obtaining tissue for vaccine production
6. Performance status (ECOG) of 0 or 1
7. Asymptomatic disease without B symptoms or severe pruritus
8. Low tumor burden as defined by the following criteria:

   * Normal lactic dehydrogenase
   * Largest tumor mass < 7 cm
   * Involvement of < 3 nodal sites with a diameter ≥ 3 cm
   * No clinically significant pleural effusion or ascites
   * Spleen size of ≤ 16 cm by CT scan
   * Circulating tumor cells < 5.0 x 109/L
   * No clinically significant organ compression
9. Adequate hematopoietic parameters:

   * Absolute neutrophil count ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Hemoglobin ≥ 10 g/dL
10. Serum creatinine ≤ 2 x upper limit of normal (ULN)
11. Total bilirubin ≤ 2 x ULN unless considered secondary to Gilbert's syndrome. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase ≤ 2 x ULN
12. Fertile patients must use effective contraception during and for 12 months after completion of therapy
13. For fertile female patients, a negative pregnancy test result at enrollment

Exclusion Criteria:

1. Active HIV, hepatitis B, hepatitis C or other active infectious process
2. Pregnant or nursing women
3. Patients with previous history of malignancy within the past 2 years except curatively treated squamous or basal cell carcinoma of the skin or curatively treated carcinoma in situ of the cervix.
4. Any medical or psychiatric condition that in the opinion of the principal investigator would compromise the patient's ability to tolerate this treatment
5. Concurrent treatment with immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall tumor response rate | Up to 2 years
  Tumor measurements will be performed at enrollment (baseline); then, tumor measurements and response assessments will occur 4 weeks after the 5th vaccination. Thereafter, tumor measurements and response assessments will occur every 3 months during the 1st year and then every 6 months during the 2nd year until relapse or disease progression, whichever occurs first.

SECONDARY OUTCOMES:
Assessment of complete and partial tumor response rates | Up to 2 years
  Tumor measurements will be performed at enrollment (baseline); then, tumor measurements and response assessments will occur 4 weeks after the 5th vaccination. Thereafter, tumor measurements and response assessments will occur every 3 months during the 1st year and then every 6 months during the 2nd year until relapse or disease progression, whichever occurs first.
Assessment of time until initiation of radiotherapy or systemic therapy | Up to 2 years
Safety evaluation will include frequency, severity, and relationship of adverse events to vaccination; vital signs (blood pressure, respiration, pulse, and temperature); and laboratory test results (including, hematology and clinical chemistry) | From the time of informed consent up to 2 years
  Safety parameters (e.g., adverse events, vital signs, and laboratory test results) will be recorded from the time patient signs informed consent, at every clinic visit during study treatment, 4 weeks after the 5th vaccination, and thereafter every 3 months during the 1st year and then every 6 months during the 2nd year.
Tests to measure tumor-specific antibody production and T cell and B cell responses to vaccination | From 8 weeks prior to the 1st vaccination to Week 19 following the 1st vaccination.
  Antibody production will be reported as increased titers of antibodies, B cells will be expressed as % B cell populations, T cell responses will be expressed as increases of tumor-specific T cells and changes in expression and quantity of cytokines (proteins that indicate changes in the immune response). Blood samples will be collected within 8 weeks prior to the 1st vaccination (baseline); within 7 days prior to the 5th vaccination; and 4 weeks after the 5th vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Brion Randolph, MD, Principal Investigator — Southeastern Regional Medical Center at Cancer Treatment Centers of America
Locations (1):
- Southeastern Regional Medical Center at CTCA, Newnan, Georgia, United States